CLINICAL TRIAL: NCT00764426
Title: Clinical Study of the Effect of Different Alcoholic and Non-Alcoholic Beverages on Markers of Inflammation
Brief Title: Alcohol, Inflammation and Atherosclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: European Research Advisory Board (Other)
Responsible Party: ERAB
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: EA 03 06
Record Dates: First submitted 2008-09-30; First posted 2008-10-02 (Estimated); Last update posted 2008-10-02 (Estimated); Status verified 2008-10

CONDITIONS: Arteriosclerosis; Myocardial Infarction
Keywords: alcoholic beverages; non-alcoholic beverages; inflammation; Serum concentration of inflammatory markers before and after intervention
MeSH Terms: conditions — Arteriosclerosis; Myocardial Infarction; Inflammation | interventions — Beer; Ethanol; Water

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- non-alcoholic beverages (Active Comparator): dealcoholised red wine, de-alcoholised beer, water
  Interventions: Drug: de-alcoholised red wine, de-alcoholised beer, water
- alcoholic beverages (Active Comparator): red wine, beer, ethanol
  Interventions: Drug: red wine, beer, ethanol

INTERVENTIONS:
Drug: red wine, beer, ethanol — Alcoholic beverages equivalent to 30g of alcohol per day for men and 20g/d for women for 3 weeks
  Arms: alcoholic beverages
Drug: de-alcoholised red wine, de-alcoholised beer, water — de-alcoholised red wine, de-alcoholised beer, water
  Arms: non-alcoholic beverages

SUMMARY:
Effect of moderate alcohol consumption in form of red wine, beer and ethanol solution and corresponding de-alcoholised beverages on immune measures.

* In healthy middle aged men and women
* In a randomized controlled cross-over trial
* Two intervention periods over 3 weeks

DETAILED DESCRIPTION:
Alcohol consumption and mortality from all causes are associated in a U-shaped manner. That means that individuals who regularly consume moderate amounts of alcohol (~1 to 2 drinks/day at maximum) on average live longer than abstainers or heavy drinkers. This is primarily through a reduced risk for fatal or non-fatal coronary heart disease events (CHD) such as myocardial infarction. In the last 10 to 15 years compelling evidence has bolstered the hypothesis that atherosclerosis is at least in part an inflammatory disease. It is also known, that alcohol influences the immune system. These facts make an impact of alcohol on the various stages of atherosclerosis via anti-inflammatory effects a reasonable assumption.

To test the effect of moderate amounts of different types of alcoholic beverages on markers of inflammation with high predictive potential for atherothrombotic complications of atherosclerosis will be examined in a cross-over short-term interventional trial. Six groups, each comprising 12 healthy individuals aged 22-56 will be included. After two weeks of abstinence from alcoholic beverages two cross-over interventional phases (each lasting 3 weeks) with red wine, beer, de-alcoholised red wine and beer of the same brand, ethanol, or water will follow. The interventions will be followed by a wash-out period of 2 weeks. Several inflammatory markers and in-vitro migration of freshly isolated monocytes will be determined before and after intervention.

ELIGIBILITY:
Inclusion Criteria:

* 20-60 years
* non-smoker
* healthy

Exclusion Criteria:

* personal or family history of dependency
* any chronic disease
* acute and chronic inflammatory processes

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2004-06

PRIMARY OUTCOMES:
Concentration of inflammatory markers including C-reactive protein | 12 weeks

SECONDARY OUTCOMES:
Ex vivo migration of monocytes | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Armin P Imhof, MD, Principal Investigator — University of Ulm, Medical Center, Ulm, Germany
Locations (1):
- University of Ulm, Medical Center, Ulm, Germany

REFERENCES:
- [Result] Imhof A, Blagieva R, Marx N, Koenig W. Drinking modulates monocyte migration in healthy subjects: a randomised intervention study of water, ethanol, red wine and beer with or without alcohol. Diab Vasc Dis Res. 2008 Mar;5(1):48-53. doi: 10.3132/dvdr.2008.009. PMID 18398813